CLINICAL TRIAL: NCT05168696
Title: The Effect of Virtual Reality Glasses Application on Anxiety and Fatigue in Women With Breast Cancer Receiving Adjuvant Chemotherapy: Pretest-Posttest Randomized Controlled Study
Brief Title: The Effect of Virtual Reality on Anxiety and Fatigue in Women With Breast Cancer Receiving Adjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Arzu USLU, RN, MS, PhD(c), Instructor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21149002
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer Female; Anxiety; Fatigue
Keywords: Virtual reality; Distraction; Anxiety; Fatigue; Nursing
MeSH Terms: conditions — Anxiety Disorders; Fatigue

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality in Women with Breast Cancer (Experimental): It is planned to pre-test, wear virtual reality glasses and post-test before chemotherapy for breast cancer women who will receive adjuvant treatment for the first time, who agree to participate in the study. This follow-up will be done 3 more times, and each cure will be followed for 4 cures. It will be ensured that the patients fill out the State Anxiety Scale and Cancer Fatigue Scale as a pre-test and post-test. After the chemotherapy infusion starts, the patient will listen and watch the relaxing beach and nature content with 360 degrees for 30 minutes with virtual reality glasses attached to the patient.
  Interventions: Other: Virtual Reality Glasses
- Standard Care in Women with Breast Cancer (No Intervention): Women with breast cancer who will receive adjuvant treatment for the first time, who agree to participate in the study, will be pre-tested before chemotherapy and a post-test will be performed 30 minutes after the start of chemotherapy treatment by the nurse. This follow-up will be done 3 more times, and each cure will be followed for 4 cures. It will be ensured that the patients fill out the State Anxiety Scale and Cancer Fatigue Scale as a pre-test and post-test.

INTERVENTIONS:
Other: Virtual Reality Glasses — Virtual Reality Glasses
  Arms: Virtual Reality in Women with Breast Cancer

SUMMARY:
It was aimed to determine the effect of virtual reality glasses application on anxiety and fatigue in women with breast cancer receiving adjuvant chemotherapy.

DETAILED DESCRIPTION:
The number of women with breast cancer worldwide is increasing day by day. Uncertainty of the efficacy of treatment, difficulty in accepting the disease, financial difficulties, insomnia, fear and anxiety about the future, concentration disorder, feeling angry, focusing on thoughts of illness and death, irregularities in work and family life, emergence of treatment Their quality of life is adversely affected due to many conditions such as worrying about side effects and loss of appetite. The disease process should be managed correctly before these symptoms related to treatment occur in patients. Anxiety and fatigue are the leading symptoms that limit the activities of daily living and significantly affect the social lives of patients receiving chemotherapy for the first time after the diagnosis of breast cancer. 46%-71% of patients diagnosed with cancer experience anxiety and 80%-90% fatigue during chemotherapy. Nurses, who are health professionals, use non-pharmacological methods as well as pharmacological methods in the prevention and management of symptoms during the chemotherapy treatment process. Non-pharmacological methods include practices such as meditation, yoga, hypnosis, prayer, relaxation techniques, daydreaming, and cognitive behavioral therapies that involve distraction. With these cognitive behavioral therapies, nurses aim to strengthen the self-care of cancer patients, increase adherence to the disease, develop effective coping methods, manage chemotherapy-related side effects, and increase hope and belief. With the method of distraction, which is frequently used from cognitive behavioral therapies, it is aimed to focus on another stimulus and to get away from negative feelings and thoughts. Recently, virtual reality application has been used frequently in the field of health for the method of distraction. Virtual reality is defined as the human computer interface that makes it feel as if it is in another universe with tools. The three-dimensional screen provides the attention of the person with the virtual reality stimuli with the motion detection system. The virtual reality application that attracts attention is preferred because it is a non-invasive intervention, has an affordable cost, and is effective in the motivation and well-being of the individual. In the meta-analysis of cancer-related symptom management, virtual reality applications, which do not require any special training, were found to increase tolerance to chemotherapy, to be effective in symptom management, to increase quality of life, and to enable acceptance of chronic disease. In the study, it was also stated that virtual reality applications were effective in reducing anxiety, depression, pain and cognitive function symptoms, although not effective in reducing fatigue, it was beneficial, and no serious side effects were reported. It is seen that the studies were designed as a single-time measurement, non-randomized research design, and a single-group pre-test-post-test. In this study, which aims to evaluate the effect of virtual reality glasses application on anxiety and fatigue in women with breast cancer receiving adjuvant chemotherapy, it is planned to increase the level of evidence of virtual reality glasses application by making multiple measurements and to evaluate fatigue with physical, emotional and cognitive sub-dimensions. In addition, this study is important in terms of increasing the awareness of oncology nurses who care for breast cancer patients about virtual reality application and integrating the method of distraction with virtual reality application into standard care. It is thought that it is useful and appropriate for the nurse to manage the distraction method with the virtual reality application, which is a non-invasive intervention, does not require specific skills, and has no serious side effects. For this purpose, it was planned to determine the effect of virtual reality glasses application on anxiety and fatigue in women with breast cancer receiving adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18 - 65
* Those who are women
* Those who were diagnosed with breast cancer for the first time and received adjuvant chemotherapy treatment
* Patients receiving the protocol with Cyclophosphamide, Doxorubicin (Adriamycin)
* Those who know that they have breast cancer
* Those with the least education level who are literate
* Those who agreed to participate in the study
* Those who speak and understand Turkish

Exclusion Criteria:

* Those receiving neoadjuvant chemotherapy treatment
* Those with metastases
* Recurrent (Recurrent) ones
* Those who use psychiatric drugs
* Those with a history of seizures
* Those with communication problems (hearing, seeing, speaking, etc.)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale | 1st cure, 2nd cure, 3rd cure, 4th cure, Each cure is given every 21 days.
  The mean anxiety scores of virtual reality glasses application in women with breast cancer receiving adjuvant chemotherapy are different from the control group. A minimum of 20 points and a maximum of 80 points are taken from the scale. The higher the score, the higher the anxiety.
Cancer Fatigue Scale | 1st cure, 2nd cure, 3rd cure, 4th cure, Each cure is given every 21 days.
  The mean fatigue scores of virtual reality glasses application in women with breast cancer receiving adjuvant chemotherapy are different from the control group. A minimum of 15 points and a maximum of 60 points are taken from the scale. The higher the score, the higher the fatigue.

SECONDARY OUTCOMES:
Cancer Fatigue Scale | 1st cure, 2nd cure, 3rd cure, 4th cure, Each cure is given every 21 days.
  The physical function sub-dimension mean scores of fatigue of virtual reality glasses application in women with breast cancer receiving adjuvant chemotherapy are different from the control group. A minimum of 7 points and a maximum of 28 points are taken from the scale. As the score increases, physical fatigue increases.
Cancer Fatigue Scale | 1st cure, 2nd cure, 3rd cure, 4th cure, Each cure is given every 21 days.
  The emotional function sub-dimension mean scores of fatigue of virtual reality glasses application in women with breast cancer receiving adjuvant chemotherapy are different from the control group. A minimum of 4 points and a maximum of 16 points are taken from the scale. Emotional fatigue increases as the score increases.
Cancer Fatigue Scale | 1st cure, 2nd cure, 3rd cure, 4th cure, Each cure is given every 21 days.
  The cognitive function sub-dimension mean scores of fatigue of virtual reality glasses application in women with breast cancer receiving adjuvant chemotherapy are different from the control group. A minimum of 4 points and a maximum of 16 points are taken from the scale. As the score increases, cognitive fatigue increases.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu USLU, RN, MS, PhD(c), Instructor, Study Director — Necmettin Erbakan University Faculty of Nursing; Selda ARSLAN, Assoc. Prof., Principal Investigator — Necmettin Erbakan University Faculty of Nursing
Locations (1):
- Necmettin Erbakan University of Nursing Faculty, Meram, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No